CLINICAL TRIAL: NCT00568009
Title: Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Sequential Cohort Study to Evaluate the Effect of SLV320 in Addition to Chronic Furosemide Treatment on Renal Function in Subjects With Congestive Heart Failure and Impaired Renal Function
Brief Title: Study to Evaluate the Effect of SLV320 in Addition to Chronic Furosemide Treatment on Renal Function in Subjects With Congestive Heart Failure and Impaired Renal Function
Status: Terminated | Type: Observational
Why Stopped: additional enrolment criteria made patients' recruitment not feasible anymore
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Kay-Christen Meyer, Solvay Pharmaceuticals
Other Study IDs: S320.2.003; 2007-000490-40
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Impaired Renal Function
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — SLV320 compound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not aplicable
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SLV320 — 1, 2.5, 5, 10 and 20 mg twice daily and placebo group. Duration of treatment 84 days

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center, sequential cohort study in subjects with congestive heart failure (CHF) and impaired renal function who are on stable furosemide treatment (³ 40 mg daily). A total of 50 subjects will be randomized to each increasing dose level of SLV320 or placebo in a sequential fashion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to85 years who gave written informed consent.
* Subjects must have a history of chronic, symptomatic, New York Heart Association (NYHA) Class II-III CHF and impaired renal function (baseline eGFR of 20 to 75 mL/min/1.73m2).
* Congestive heart failure should have been diagnosed at least 3 months before Visit 1 (Day 1) and the subjects should be on chronic treatment with furosemide (40 mg daily) for at least 3 weeks before Visit 1 (Day 1).
* Subjects must be on stable doses of their individually optimized medication regimen for at least 4 weeks before Visit 1 (Day 1).

Exclusion Criteria:

* Any history of a convulsive disorder or pre-convulsive state and any risk for a convulsive disorder or pre-convulsive state (for example any past brain trauma, abuse of alcohol) will lead to an exclusion from the study.
* Females of childbearing potential not using specified contraception, subjects with malignant tumors with a short life expectancy, subjects with known severe reactions to drugs and subjects with bilateral renal artery stenosis will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Congestive Heart Failure, Impaired Renal Function
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Cystatine C | 3 months

SECONDARY OUTCOMES:
Sodium in urine | 3 months
Estimated glomerular filtration rate | 3 months
Clinical global impression | 3 months
Body weight | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (72):
- United States (10):
  - Site 96, Whittier, California
  - Site 95, Largo, Florida
  - Site 90, Miami, Florida
  - Site 88, Atlanta, Georgia
  - Site 92, Covington, Georgia
  - Site 106, Melrose Park, Illinois
  - Site 87, Hagerstown, Maryland
  - Site 94, Springfield Gardens, New York
  - Site 89, Dallas, Texas
  - Site 97, San Antonio, Texas
- Argentina (11):
  - Site 11, Bahía Blanca
  - Site 2, Bahía Blanca
  - Site 101, Capital Federal
  - Site 6, Coronel Suárez
  - Site 1, Corrientes
  - Site 5, La Plata
  - Site 104, Mar del Plata
  - Site 102, Salta
  - Site 105, San Luis
  - Site 4, San Martín
  - Site 8, Santa Fe
- Belgium (3):
  - Site 14, Antwerp
  - Site 15, Ghent
  - Site 12, Huy
- Czechia (8):
  - Site 22, Brno
  - Site 16, Jindřichův Hradec
  - Site 19, Kroměříž
  - Site 20, Prague
  - Site 21, Prague
  - Site 17, Semily
  - Site 18, Slaný
  - Site 23, Teplice
- Germany (3):
  - Site 24, Bad Nauheim
  - Site 28, Berlin
  - Site 26, Dortmund
- Poland (11):
  - Site 50, Bydgoszcz
  - Site 47, Lublin
  - Site 49, Płock
  - Site 57, Skierniewice
  - Site 54, Torun
  - Site 48, Warsaw
  - Site 52, Warsaw
  - Site 53, Warsaw
  - Site 56, Warsaw
  - Site 55, Wroclaw
  - Site 51, Zielona Góra
- Russia (7):
  - Site 58, Moscow
  - Site 61, Moscow
  - Site 62, Moscow
  - Site 63, Moscow
  - Site 64, Moscow
  - Site 60, Saint Petersburg
  - Site 59, Samara
- Serbia and Montenegro (6):
  - Site 65, Belgrade
  - Site 66, Belgrade
  - Site 69, Belgrade
  - Site 68, Niska Banja
  - Site 67, Sremska Kamenica
  - Site 70, Zemun
- South Africa (7):
  - Site 72, Belville
  - Site 75, Belville
  - Site 76, Bloemfontein
  - Site 98, Durban
  - Site 73, Kempton Park
  - Site 71, Somerset West
  - Site 74, Worcester
- Spain (6):
  - Site 78, Barcelona
  - Site 83, Barcelona
  - Site 79, Madrid
  - Site 77, Málaga
  - Site 82, Santander
  - Site 80, Valencia